CLINICAL TRIAL: NCT00524303
Title: Phase II Randomized Trial of Neoadjuvant Trastuzumab and/or Lapatinib Plus Chemotherapy (Sequential FEC75 and Paclitaxel) in Women With ErbB2- (HER2/Neu-) Overexpressing Invasive Breast Cancer
Brief Title: Lapatinib +/- Trastuzumab In Addition To Standard Neoadjuvant Breast Cancer Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPT109096
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2011-08-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-03

CONDITIONS: Neoplasms, Breast
Keywords: ErbB2 Overexpressing; ErbB2 Positive; Lapatinib; Invasive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Active Comparator): Trastuzumab alone for 2 weeks then in combination with FEC75 for 4 (21 Day) cycles and Paclitaxel for 4 (21 day) cycles then continued trastuzumab until time of definitive surgery
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: FEC75
- Arm 2 (Experimental): Lapatinib alone for 2 weeks then in combination with FEC75 for 4 (21 Day) cycles followed by Paclitaxel for 4 (21 day) cycles then continued lapatinib until time of definitive surgery
  Interventions: Drug: Paclitaxel; Drug: FEC75; Drug: Lapatinib
- Arm 3 (Experimental): Trastuzumab + Lapatinib for 2 weeks then added FEC75 for 4 (21 Day) cycles followed by Paclitaxel for 4 (21 day) cycles then continued trastuzumab + lapatinib until time of definitive surgery
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: FEC75; Drug: Lapatinib

INTERVENTIONS:
Drug: Trastuzumab — 4mg/kg IV loading dose followed by 2mg/kg IV weekly
  Arms: Arm 1; Arm 3
Drug: Paclitaxel — 80mg/m2 IV weekly for 4 (21 day) cycles
Drug: FEC75 — 5FU 500mg/m2 + Epirubicin 75 mg/m2 + cyclophosphamide 500 mg/m2 IV on day 1 of 4 (21 day) cycles
Drug: Lapatinib — 1250 mg oral daily dose in arm 2, 750 mg oral daily dose for FEC cycles and then 1000 mg oral daily dose during the Paclitaxel cycles in arm 3
  Arms: Arm 2; Arm 3

SUMMARY:
This study will examine safety and efficacy of Lapatinib in combination with a standard neoadjuvant chemotherapy including 5FU, Epirubicin, Cyclophosphamide and Paclitaxel. Tumor tissue will be obtained at 3 timepoints (optional 4th) to evaluate tumor response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an informed consent form (ICF) and a Patient Authorization Form (HIPAA).
* Have histologically or cytologically confirmed ErbB2- (HER2/neu-) overexpressing invasive breast cancer (T2-4, N0-2).
* ErbB2 overexpressing breast cancer, defined as one of the following definitions:
* 3+ staining by immunohistochemistry (IHC),
* a fluorescent in situ hybridization (FISH) result of more than six HER2 gene copies per nucleus
* a FISH ratio of more than 2.2.
* Have either measurable or evaluable disease.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1 (Refer to Section 11.4).
* Have LVEF within the institutional range of normal as measured by either echocardiogram (ECHO) or MUGA scans. The same modality must be used consistently throughout the study.
* Be deemed able to tolerate 8 cycles of preoperative chemotherapy, including 4 cycles with an anthracycline (epirubicin).
* Must be willing to undergo 2 mandatory core biopsies (4 passes each) after diagnosis to obtain tissue for biologic expression profiling. Any subject with clinically palpable residual disease may undergo an optional third biopsy to allow identification of presumed pathways of resistance to therapy. This information might be useful in providing the subject with options for other targeted therapies if definitive surgery confirms residual disease. Definitive local therapy with surgery and radiation therapy as indicated will be performed after completion of 12 weeks of paclitaxel-based chemotherapy.
* Are able to swallow and retain oral medication (intact pill).
* Are able to complete all screening assessments as outlined in the protocol.
* Have adequate organ function as defined in Table 4:

Table 1 Baseline Laboratory Values

Hematologic:

ANC (absolute neutrophil count) >1.5 x 109/L hemoglobin >9 g/dL platelets >75 x 109/L

Hepatic:

albumin >2.5 g/dL serum bilirubin <1.25 x ULN AST / ALT <3 x ULN if no documented liver metastases AST / ALT <3 x ULN with documented liver metastases

Renal:

serum creatinine <2.0 mg/dL

* OR - calculated creatinine clearance >40 mL/min
* Are subjects aged >18 years with any menopausal status:

Non-child-bearing potential (i.e., women with functioning ovaries who have a current documented tubal ligation or hysterectomy, or women who are postmenopausal)

Child-bearing potential (i.e., women with functioning ovaries and no documented impairment of oviductal or uterine function that would cause sterility.) This category includes women with oligomenorrhea (severe), women who are perimenopausal, and young women who have begun to menstruate. These subjects must have a negative serum pregnancy test at screening and agree to one of the following:

Complete abstinence from intercourse from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of study medication; or Consistent and correct use of one of the following acceptable methods of birth control: male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject; any intrauterine device (IUD) with a documented failure rate of less than 1% per year; oral contraceptives (either combined or progestogen only) where not contraindicated for this subject population or per local practice.; or barrier methods, including diaphragm or condom with a spermicide.

Please note that breast cancer subjects on this trial cannot receive injectable levonorgestrel or injectable progestogen due to the potential for an adverse effect of anti-hormonal therapies on chemotherapy administered for breast cancer [Albain, 2002]. Progestogen may also affect the proliferative rate of endocrine-responsive tumors.

Exclusion Criteria:

* Have received any prior chemotherapy.
* Had prior therapy with an ErbB1 and/or ErbB2 inhibitor.
* Are receiving concurrent anti-cancer therapy (chemotherapy, immunotherapy, and biologic therapy) while taking study medication.
* Have malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel. Women with ulcerative colitis are also excluded.
* Have a concurrent disease or condition that would make the woman inappropriate for study participation, or any serious medical disorder that would interfere with the woman's safety.
* Have an active or uncontrolled infection.
* Have dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.
* Have active cardiac disease, defined as one or more of the following:

History of uncontrolled or symptomatic angina History of arrhythmias requiring medications, or clinically significant Myocardial infarction <6 months from study entry Uncontrolled or symptomatic congestive heart failure Ejection fraction below the institutional normal limit Any other cardiac condition, which in the opinion of the treating physician, would make this protocol unreasonably hazardous for the patient

* Are pregnant or breastfeeding.
* Have received concurrent treatment with an investigational agent or participate in another clinical trial.
* Have received concurrent treatment with prohibited medications (refer to Section 5.8.2 for details on prohibited medications).
* Have used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication.
* Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to any of the agents used in this study or their excipients.
* Are receiving therapeutic anti-coagulation therapy (i.e. warfarin, heparin).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (21):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Hudson, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Bedford, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lewisville, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Yakima, Washington

REFERENCES:
- [Derived] O'Shea J, Cremona M, Morgan C, Milewska M, Holmes F, Espina V, Liotta L, O'Shaughnessy J, Toomey S, Madden SF, Carr A, Elster N, Hennessy BT, Eustace AJ. A preclinical evaluation of the MEK inhibitor refametinib in HER2-positive breast cancer cell lines including those with acquired resistance to trastuzumab or lapatinib. Oncotarget. 2017 Jul 22;8(49):85120-85135. doi: 10.18632/oncotarget.19461. eCollection 2017 Oct 17. PMID 29156708
- [Derived] Holmes FA, Espina V, Liotta LA, Nagarwala YM, Danso M, McIntyre KJ, Osborne CR, Anderson T, Krekow L, Blum JL, Pippen J, Florance A, Mahoney J, O'Shaughnessy JA. Pathologic complete response after preoperative anti-HER2 therapy correlates with alterations in PTEN, FOXO, phosphorylated Stat5, and autophagy protein signaling. BMC Res Notes. 2013 Dec 5;6:507. doi: 10.1186/1756-0500-6-507. PMID 24304724

RESULTS

PARTICIPANT FLOW:
Groups:
- Trastuzumab: Participants received trastuzumab alone (a loading dose of 4 milligrams [mg]/kilogram [kg] on Day 1, followed by a dose of 2 mg/kg on Day 1 of Week 2 and weekly thereafter). Participants were treated with trastuzumab in a 2-week run-in period. On Day 14, a second core needle biopsy was performed, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each (1 cycle=3 weeks): FEC75 (5-fluorouracil [5-FU] 500 mg/meters squared [m^2], epirubicin 75 mg/m^2, cyclophosphamide 500 mg/m^2 x 4 cycles on Day 1), then paclitaxel (80 mg/m^2 x 4 cycles on Day 1, Day 8, and Day 15) in combination with trastuzumab.
- Lapatinib: Participants received lapatinib alone (1250 mg orally [PO] once daily [QD]). Participants were treated with lapatinib in a 2-week run-in period. On Day 14, a second core needle biopsy was performed, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each (1 cycle=3 weeks): FEC75 (5-FU 500 mg/m^2, epirubicin 75 mg/m^2, cyclophosphamide 500 mg/m^2 x 4 cycles on Day 1), then paclitaxel (80 mg/m^2 x 4 cycles on Day 1, Day 8, and Day 15) in combination with lapatinib.
- Trastuzumab+Lapatinib: Participants received trastuzumab (given as in Arm 1) and lapatinib (750/1000 mg PO QD). Participants were treated with these medications in a 2-week run-in period. On Day 14, a second core needle biopsy was performed, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each (1 cycle=3 weeks): FEC75 (5-FU 500 mg/m^2, epirubicin 75 mg/m^2, cyclophosphamide 500 mg/m^2 x 4 cycles on Day 1), then paclitaxel (80 mg/m^2 x 4 cycles on Day 1, Day 8, and Day 15) in combination with trastuzumab+lapatinib.
Period: Overall Study
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Started | 33 | 34 | 33
Completed | 21 | 24 | 15
Not Completed | 12 | 10 | 18
Not completed — Lost to Follow-up | 6 | 0 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0 | 4
Not completed — Death | 0 | 2 | 3
Not completed — Adverse Event | 1 | 2 | 3
Not completed — Did not Complete Study Dosing | 1 | 0 | 0
Not completed — Worsening Peripheral Neuropathy | 1 | 0 | 0
Not completed — Disease Progression | 0 | 4 | 1
Not completed — Disease Recurrence | 0 | 1 | 0
Not completed — Sponsor Request | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Completed 5 years | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib | Total
Number analyzed (Participants) | 33 | 34 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (10.90) | 50.8 (8.76) | 49.2 (10.47) | 50.4 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 33 | 100
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African heritage | 8 | 1 | 2 | 11
  American Indian or Alaska native | 0 | 0 | 1 | 1
  Asian - Central/South Asian heritage | 0 | 1 | 0 | 1
  Asian - East Asian heritage | 0 | 1 | 0 | 1
  Asian - South East Asian heritage | 0 | 2 | 1 | 3
  White - Arabic/North African heritage | 0 | 1 | 0 | 1
  White - White/Caucasian/European heritage | 25 | 27 | 29 | 81
  Mixed race | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Pathological Complete Response (pCR) After 26 Weeks of Therapy
Description: A pCR in the breast was defined as no pathologic evidence of invasive disease (residual ductal carcinoma in situ [DCIS] or lobular carcinoma in situ [LCIS] was allowed). A pCR in the axillary lymph node(s) was defined as no evidence of breast cancer cells in the lymph node (including subcapsular sinus). Overall pCR was defined as the sum of pCR in the breast and pCR in the lymph nodes. 26 weeks of therapy comprised the 2-week run-in phase, 12 weeks of treatment with FEC, and 12 weeks of treatment with Paclitaxel.
Time Frame: Week 26
Population: Intent-to-Treat-Evaluable (ITT-E) Population: ITT participants with evaluable tumor responses who had been >=75% compliant to 5-fluorouracil (5-FU) 500 mg/m^2, epirubicin 75 mg/m^2, cyclophosphamide 500 mg/m^2 (FEC75) and paclitaxel 80 mg/m^2 and had undergone surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Number analyzed (Participants) | 26 | 29 | 23
percentage of participants | 54.0 | 45.0 | 74.0
Statistical Analysis 1: Comparison: Trastuzumab vs Lapatinib; Test type: Superiority or Other; Percent difference = -9, 95% CI 2-sided [-38.1 to 17.9] — Approximate 95% confidence interval for the difference in response rates between the trastuzumab arm and the lapatinib arm was calculated
Statistical Analysis 2: Comparison: Trastuzumab vs Trastuzumab+Lapatinib; Test type: Superiority or Other; Percent difference = 20, 95% CI 2-sided [-8.0 to 49.4] — Approximate 95% confidence interval for the difference in response rates between the transtuzumab arm and the transtuzumab + lapatinib arm was calculated

2. Secondary Outcome: Percentage of Participants With Clinical Complete Response (cCR) at 26 Weeks or at End of Treatment (EOT) or Early Withdrawal
Description: cCR was defined as the percentage of participants achieving either a Complete Response (CR) or a Partial Response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR was defined as the disappearance of all target lesions, and PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Week 26 or EOT or Early withdrawal
Population: ITT Population: all randomized participants regardless of whether they had received any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Number analyzed (Participants) | 33 | 34 | 33
percentage of participants | 61.0 | 68.0 | 61.0
Statistical Analysis 1: Comparison: Trastuzumab vs Lapatinib; Test type: Superiority or Other; p = 0.627, Fisher Exact; Percent Difference = 7, 95% CI 2-sided [-17.8 to 32.5] — Approximate 95% confidence interval for the difference in response rates between the transtuzumab arm and the lapatinib arm was calculated
Statistical Analysis 2: Comparison: Trastuzumab vs Trastuzumab+Lapatinib; Test type: Superiority or Other; p = 1.000, Fisher Exact; Percent Difference = 0, 95% CI 2-sided [-25.1 to 25.1] — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: Percentage of Participants (Par.) With Disease-free Survival (DFS) at the End of 5 Years From Randomization
Description: Percentage is the Kaplan Meier estimate of DFS. DFS is time from randomization until disease recurrence (contralateral breast cancer; second primary cancer; progression during neo-adjuvant treatment; or death from any cause). Par. who experienced progression during treatment and were withdrawn were considered to have a DFS event at withdrawal.
Time Frame: From first dose date until disease progression, assessed up to a maximum of 5 years
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Number analyzed (Participants) | 33 | 34 | 33
Percentage | 90 [72 to 97] | 67 [47 to 80] | 66 [44 to 82]

4. Secondary Outcome: Number of Participants With the Indicated Electrocardiogram (ECG) Status at Baseline and at EOT or Early Withdrawal
Description: 12-lead ECGs were performed, and participants were classified as having normal ECG, abnormal- not clinically significant (NCS) ECG, and abnormal-clinically significant (CS) ECG per investigator opinion and reported result.
Time Frame: Baseline and EOT (up to Week 26) or Early withdrawal
Population: Safety Population: all randomized participants (par) who received at least one dose of investigational product, based on actual treatment received if this differed from that to which par was randomized. Not all par were analyzed: some par were randomized to an arm they did not want or par were randomized in error (eligibility criteria weren't met).
Measure: Number; unit: participants
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Number analyzed (Participants) | 28 | 32 | 30
participants
  Baseline, Normal, n= 28, 32, 30 | 18 | 23 | 23
  Baseline, Abnormal-NCS, n= 28, 32, 30 | 10 | 8 | 7
  Baseline, Abnormal-CS, n= 28, 32, 30 | 0 | 1 | 0
  EOT/early withdrawal, Normal, n= 16, 21, 16 | 10 | 12 | 12
  EOT/early withdrawal, Abnormal-NCS, n= 16, 21, 16 | 6 | 8 | 4
  EOT/early withdrawal, Abnormal-CS, n= 16, 21, 16 | 0 | 1 | 0

5. Secondary Outcome: Cumulative Number of Participants With at Least One Decrease of More Than or Equal to 20% in Left Ventricular Ejection Fraction (LVEF) at the Indicated Time Points Compared to LVEF at Baseline
Description: LVEF is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction and is used to determine cardiac function. LVEF was measured by performing echocardiogram (ECHO). If ECHO could not be performed or if the investigator believed that it was not conclusive to evaluate LVEF, then a multigated acquisition (MUGA) scan was performed.
Time Frame: Weeks 3, 9, and 15; EOT or early withdrawal; and 3- and 6-month survival follow-up after last chemotherapy course
Population: Safety Population. Not all participants in the Safety Population were analyzed: some participants were randomized to an arm they did not want or participants were randomized in error (eligibility criteria weren't met).
Measure: Number; unit: participants
Groups:
- Trastuzumab: Participants received trastuzumab alone (a loading dose of 4 milligrams (mg)/kilogram (kg) on Day 1, followed by a dose of 2 mg/kg on Day 1 of Week 2 and weekly thereafter. Participants were treated with trastuzumab in a 2-week run-in period. On Day 14, a second core needle biopsy was performed, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each (1 cycle=3 weeks): FEC75 (5-fluorouracil [5-FU] 500 mg/meters squared [m^2], epirubicin 75 mg/m^2, cyclophosphamide 500 mg/m^2 x 4 cycles on Day 1), then paclitaxel 80 mg/m^2 x 4 cycles on Day 1, Day 8, and Day 15) in combination with trastuzumab.
- Lapatinib: Participants received lapatinib alone (1250 mg orally [PO] once daily [QD]). Participants were treated with lapatinib in a 2-week run-in period. On Day 14, a second core needle biopsy was performed, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each (1 cycle=3 weeks): FEC75 (5-FU 500 mg/m^2, epirubicin 75 mg/m^2, cyclophosphamide 500 mg/m^2 x 4 cycles on Day 1), then paclitaxel 80 mg/m^2 x 4 cycles on Day 1, Day 8, and Day 15) in combination with lapatinib.
- Trastuzumab+Lapatinib: Participants received trastuzumab (given as in Arm 1) and lapatinib (750/1000 mg PO QD). Participants were treated with these medications in a 2-week run-in period. On Day 14, a second core needle biopsy was performed, followed by initiation of chemotherapy with 2 combination regimens of 4 cycles each (1 cycle=3 weeks): FEC75 (5-FU 500 mg/m^2, epirubicin 75 mg/m^2, cyclophosphamide 500 mg/m^2 x 4 cycles on Day 1), then paclitaxel 80 mg/m^2 x 4 cycles on Day 1, Day 8, and Day 15) in combination with trastuzumab+lapatinib.
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Number analyzed (Participants) | 32 | 34 | 31
participants
  Week 3, n= 30, 31, 26 | 1 | 0 | 1
  Week 9, n= 30, 32, 27 | 1 | 0 | 1
  Week 15, n= 31, 34, 28 | 1 | 2 | 2
  Early withdrawal/EOT, n= 31, 34, 28 | 1 | 4 | 2
  3-month survival follow-up, n= 31, 34, 28 | 2 | 4 | 3
  6-month survival follow-up, n= 31, 34, 28 | 4 | 4 | 4

6. Other Pre Specified Outcome: Mean Intra-tumoral Expression of the Indicated Proteins at Baseline and Day 14
Description: Expression (exp) of biomarker proteins (prot) were analyzed to determine if individual prot levels either in the Baseline or Day 14 breast tumor biopsy specimen correlated with breast pCR. A biomarker indicates a change in exp or state of a prot that correlates with the risk or disease progression, or with the susceptibility of the disease to a given treatment. Biomarkers are characteristic biological properties that can be detected and measured in parts of the body like blood or tissue. pCR=yes: participants (par.) had breast pCR. pCR=no: par. did not have breast pCR. Prot exp values are represented as normalized, scaled values; the unit of measurement is unit-less. Raw exp values were processed as follows: background subtraction of the raw exp value, then that value divided by beta-acting exp to normalize the exp value. A Standard Z score was calculated to scale the exp value.
Time Frame: Tumor core biopsy taken at Baseline and Treatment Day 14
Population: ITT-E Population. Only those participants with matched pairs of biopsy samples for analysis at Baseline and on Day 14 were analyzed.
Measure: Mean (Standard Deviation); unit: : normalized relative expression level
Arm/Group | Trastuzumab | Lapatinib
Number analyzed (Participants) | 11 | 9
: normalized relative expression level
  Baseline, EGFR_Tyr1068; pCR=yes, n=0, 4 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | -0.70 (0.47)
  Baseline, Baseline, EGFR_Tyr1068; pCR=no, n=0, 11 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | 0.05 (0.55)
  Post Baseline, EGFR_Tyr1068; pCR=yes, n=9, 0 | 0.65 (1.02) | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm.
  Post Baseline, EGFR_Tyr1068; pCR=no, n=6, 0 | -0.26 (0.56) | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm.
  Day 14, pSTAT5; pCR=yes, n=11, 6 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm.
  Day 14, pSTAT5; pCR=no, n=9, 11 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm.
  Post Baseline, PI3K; pCR=yes, n=0, 5 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | 0.46 (0.73)
  Post Baseline, PI3K; pCR=no, n=0, 10 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | -0.53 (0.67)
  Post Baseline, LC3B; pCR=yes, n=0, 5 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | 0.68 (0.81)
  Post Baseline, LC3B; pCR=no, n=0, 10 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | -0.43 (0.75)
  Post Baseline, MMP9; pCR=yes, n=0, 5 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | 0.71 (0.34)
  Post Baseline, MMP9; pCR=no, n=0, 5 | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm. | -0.48 (0.48)
  Post Baseline, GSK3_a_b_Tyr279_216; pCR=yes, n=8,0 | 0.26 (0.82) | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm.
  Post Baseline, GSK3_a_b_Tyr279_216; pCR=no, n=5,0 | -0.86 (0.67) | NA (NA) — This protein was not significantly expressed at this time point in this treatment arm.

7. Other Pre Specified Outcome: Cancer Stem Cells and the Correlation to Response/Non-response to Treatment
Description: Stem cell data were of poor quality and thus could not be analyzed. Increases or decreases in cancer stem cells and how the changes correlated with response/non-response to treatment were to have been assessed.
Time Frame: Tumor core biopsy taken at Baseline and Treatment Day 14
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Number analyzed (Participants) | 0 | 0 | 0

8. Other Pre Specified Outcome: Transcriptional Profiling of Total RNA and the Correlation to Response/Non-response to Treatment
Description: Transcriptional data were of poor quality and thus could not be analyzed. Gene pathways that correlate with response/non-response to treatment were to have been evaluated. The unit of measure is unit less; however, the processed values would be considered normalized relative expression level.
Time Frame: Tumor core biopsy taken at Baseline and Treatment Day 14
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: In the Safety Population, serious and non-serious adverse events were collected from all randomized participants who received at least one dose of investigational product and was based on the actual treatment received if this differed from that to which the participant was randomized.
Arm/Group | Trastuzumab | Lapatinib | Trastuzumab+Lapatinib
Serious Adverse Events (participants affected / at risk) | 7/32 | 7/34 | 8/31
Other Adverse Events (participants affected / at risk) | 31/32 | 34/34 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=32) | Lapatinib (N=34) | Trastuzumab+Lapatinib (N=31)
Febrile nuetropenia (Blood and lymphatic system disorders) | 3 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cellilitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 3 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Dysponea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=32) | Lapatinib (N=34) | Trastuzumab+Lapatinib (N=31)
Nausea (Gastrointestinal disorders) | 26 | 26 | 26
Diarrhoea (Gastrointestinal disorders) | 17 | 29 | 31
Fatigue (General disorders) | 22 | 24 | 24
Rash (Skin and subcutaneous tissue disorders) | 14 | 28 | 26
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 24 | 18
Neuropathy peripheral (Nervous system disorders) | 15 | 19 | 14
Neutropenia (Blood and lymphatic system disorders) | 13 | 12 | 15
Anemia (Blood and lymphatic system disorders) | 10 | 12 | 12
Vomiting (Gastrointestinal disorders) | 7 | 15 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 10
Constipation (Gastrointestinal disorders) | 12 | 8 | 6
Dysgeusia (Nervous system disorders) | 4 | 10 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 10 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 10 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 11 | 6
Nail disorder (Skin and subcutaneous tissue disorders) | 4 | 10 | 8
Oedema peripheral (General disorders) | 5 | 10 | 7
Headache (Nervous system disorders) | 8 | 6 | 7
Mucosal inflammation (General disorders) | 6 | 7 | 8
Decreased appetite (Metabolism and nutrition disorders) | 5 | 7 | 7
Stomatitis (Gastrointestinal disorders) | 5 | 7 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 6 | 5 | 7
Pyrexia (General disorders) | 3 | 6 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 7
Insomnia (Psychiatric disorders) | 5 | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7 | 6
Abdominal pain (Gastrointestinal disorders) | 5 | 6 | 3
Anxiety (Psychiatric disorders) | 4 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3 | 5
Urinary tract infection (Infections and infestations) | 4 | 5 | 5
Pain (General disorders) | 3 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 3 | 5
Leukopenia (Blood and lymphatic system disorders) | 3 | 4 | 5
Depression (Psychiatric disorders) | 5 | 5 | 1
Haemoglobin decreased (Investigations) | 1 | 6 | 4
Dizziness (Nervous system disorders) | 3 | 5 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 4
Neutrophil count decreased (Investigations) | 2 | 4 | 3
Alanine aminotransferase increased (Investigations) | 1 | 3 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 4
Breast pain (Reproductive system and breast disorders) | 1 | 3 | 4
Dysuria (Renal and urinary disorders) | 4 | 3 | 1
Hot flush (Vascular disorders) | 4 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 3
Weight decreased (Investigations) | 0 | 3 | 5
Asthenia (General disorders) | 4 | 2 | 3
Catheter site pain (General disorders) | 5 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Chills (General disorders) | 5 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2
Oral pain (Gastrointestinal disorders) | 1 | 1 | 4
Pruritus genralised (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Rhinitis (Infections and infestations) | 2 | 3 | 1
Syncope (Nervous system disorders) | 1 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 3 | 1
Hypertension (Vascular disorders) | 1 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 2
Lacrimation increased (Eye disorders) | 3 | 0 | 2
Nasopharyngitis (Infections and infestations) | 3 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 4 | 0
Platelet count decreased (Investigations) | 1 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 2 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Vision blurred (Eye disorders) | 1 | 2 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 0
Blood lactate dehygrogenase increased (Investigations) | 1 | 1 | 2
Chest discomfort (General disorders) | 2 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2
Herpes zoster (Infections and infestations) | 1 | 1 | 2
Localised infection (Infections and infestations) | 0 | 2 | 2
Memory impairment (Nervous system disorders) | 1 | 2 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Seasonal allergy (Immune system disorders) | 1 | 2 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 1 | 1
White blood cell count decreased (Investigations) | 1 | 3 | 0
Body temperature increased (Investigations) | 3 | 0 | 0
Candidiasis (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Palpitations (Cardiac disorders) | 1 | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Tremor (Nervous system disorders) | 1 | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 0 | 1
Alanine aminotranferase decreased (Investigations) | 0 | 2 | 0
Axillary pain (General disorders) | 0 | 0 | 2
Catheter site related reaction (General disorders) | 0 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dysponoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Eye irritation (Eye disorders) | 0 | 2 | 0
Face oedema (General disorders) | 0 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.